CLINICAL TRIAL: NCT00898326
Title: Analysis of Biopsy Results at 36 Months After Permanent I-125 Implantation Therapy Plus LHRH-agonist Therapy for Patients With Untreated Intermediate Prostate Cancer.
Brief Title: PSA Levels and Biopsy Samples After Implant Radiation and Hormone Therapy in Patients With Stage I or Stage II Prostate Cancer
Acronym: SHIP36B
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Jikei University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: JUSMH-TRIGU0709; CDR0000593698 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Biopsy 36 month after breacchytherapy: Biopsy 36 month after breacchytherapy on protocol JUSMH-BRI-GU05-01.
  Interventions: Other: biopsy

INTERVENTIONS:
Other: biopsy — Conduct prostatic needle biopsy at 36-39 months-after brachy therapy. Basic method is by transectal ultra-sound-guided systematic biopsy,; systematic sextant biopsy which involves samples from both seminal vesicles is adopted as much as possible.

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with prostate cancer after receiving implant radiation therapy and luteinizing hormone-releasing hormone agonist may help doctors identify biomarkers related to cancer and help doctors predict how patients will respond to treatment.

PURPOSE: This laboratory study is looking at PSA levels and biopsy samples after undergoing implant radiation therapy and luteinizing hormone-releasing hormone agonist therapy in patients with stage I or stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To analyze biopsy results at 36 months after permanent iodine I 125 implantation therapy and luteinizing hormone-releasing hormone (LHRH) agonist therapy for patients with untreated intermediate-risk prostate cancer.

OUTLINE: Patients received luteinizing hormone releasing-hormone (LHRH) agonist therapy and permanent iodine I 125 implantation on protocol JUSMH-BRI-GU05-01.

Patients undergo blood sample collection and tissue biopsy for biomarker/laboratory analysis at 36 months after receiving brachytherapy and releasing-hormone agonist therapy. PSA levels and biopsy results are compared.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed prostate cancer

  * Previously untreated disease prior to participation on protocol JUSMH-BRI-GU05-01
* Intermediate-risk disease as defined by the following:

  * Clinical stage < T2c
  * Prostate-specific antigen (PSA) ≤ 20 ng/mL
  * Gleason score < 8
* Previously enrolled on protocol JUSMH-BRI-GU05-01

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 3 months
* WBC ≥ 2,000/μL
* Hemoglobin ≥ 10.0 g/dL
* Platelet count ≥ 100,000/μL
* Serum creatine level ≤ 2.0 mg/dL
* ALT and AST ≤ 100 IU/L
* No other cancer requiring treatment
* No poorly controlled hypertension (i.e., diastolic blood pressure ≥ 120 mm Hg)
* No severe psychiatric disorders, including schizophrenia or dementia
* No poorly controlled diabetes
* Considered appropriate for study participation, as determined by the Principal Investigator or Clinical Investigator

PRIOR CONCURRENT THERAPY:

* No prior drugs for benign prostatic hyperplasia (other than antiandrogen therapy)
* No prior surgery for prostate cancer
* No concurrent steroid drugs (except for ointment)
* No other concurrent antiandrogen therapy

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously enrolled on protocol JUSMH-BRI-GU05-01 and 36 month after treatement of brachytherapy.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of PSA levels and biopsy results at 36 months months | 36-39 month after PI-125
  Compare biobsy results and PSA revels at baseline vs. 36 months after brachytherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Shin Egawa, MD, PhD, Principal Investigator — Jikei University School of Medicine
Locations (1):
- Jikei University School of Medicine Hospital, Tokyo, Japan

REFERENCES:
- [Result] Miki K, Kiba T, Sasaki H, Kido M, Aoki M, Takahashi H, Miyakoda K, Dokiya T, Yamanaka H, Fukushima M, Egawa S. Transperineal prostate brachytherapy, using I-125 seed with or without adjuvant androgen deprivation, in patients with intermediate-risk prostate cancer: study protocol for a phase III, multicenter, randomized, controlled trial. BMC Cancer. 2010 Oct 21;10:572. doi: 10.1186/1471-2407-10-572. PMID 20964826